CLINICAL TRIAL: NCT02589002
Title: Effects of Sucralose on Insulin Sensitivity, Pancreatic Response and Appetite Regulating Hormones
Brief Title: Effects of Sucralose on Glucose Metabolism
Acronym: Sucralose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1544
Record Dates: First submitted 2015-10-15; First posted 2015-10-28 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2016-08

CONDITIONS: Glucose Metabolism Disorders
Keywords: sucralose; insulin sensitivity; beta-cell response; appetite regulating hormone
MeSH Terms: conditions — Glucose Metabolism Disorders; Insulin Resistance | interventions — trichlorosucrose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sucralose (Experimental): Ingestion of 15% of the ADI of sucralose daily during two weeks
  Interventions: Other: Sucralose
- Control (No Intervention): Absence of sucralose ingestion

INTERVENTIONS:
Other: Sucralose
  Other Names: Non-nutritive sweetener
  Arms: Sucralose

SUMMARY:
In this study the effects of sucralose on insulin sensitivity, beta-cell response and appetite regulating hormones will be evaluated.

DETAILED DESCRIPTION:
The consumption of non-nutritive sweeteners has a high prevalence. The effect of non-nutritive sweeteners in both beta-cell function and insulin resistance it is unknown.

Previous studies performed in animal models and humans with diverse characteristics have shown variable effects of different non-nutritive sweeteners in variables related to glucose metabolism.

Due to the high consumption of non-nutritive sweeteners it is relevant to know its effect in beta cell-function and insulin sensitivity.

In this study the effects of sucralose, a non-nutritive sweetener that is highly consumed in the population, on insulin sensitivity and beta-cell function will be evaluated.

54 participants with normal glucose tolerance, normal weight, and without chronic diseases with a low consumption of non-nutritive sweeteners will be included. The participants will be randomly assigned to consume sucralose or to a control group.

During the first visit an oral glucose tolerance test with 75 g of glucose will be performed. Fasting and 2-hour glucose will be measured in order to rule-out diabetes, abnormal fasting glucose, or glucose intolerance.

During the second visit a three-hour IV glucose tolerance test will be performed administering 0.3 g/kg of glucose and insulin 0.03 U/kg. Samples will be taken following the minimal model described by Bergman.

After this visit, the group assigned to receive sucralose will ingest 15% of the adequate daily intake (ADI) of sucralose and the control group will abstain of any non-nutritive sweetener consumption during 14 days. At the end of this period a third visit to repeat the IV glucose tolerance test will be performed.

Samples will be analyzed measuring glucose and insulin concentrations to evaluate acute insulin response (AIR), glucose effectiveness (SG), first phase pancreatic response (ф1), and second phase pancreatic response (ф2). In addition, hormones involved in appetite and satiety (leptin, ghrelin, and peptide tyrosine tyrosine) will be quantified at the beginning and end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* both genders
* age between 18 and 55 years
* body mass index ≥18.5 and <25 kg/m2
* low consumption of non-nutritive sweeteners

Exclusion Criteria:

* diabetes or glucose intolerance
* consumption of medications affecting insulin sensitivity (metformin, steroids, hormone replacement therapy, contraceptives)
* intestinal disease such as malabsorption or previous intestinal resection
* history of bariatric surgery
* pregnancy or lactation
* weight loss greater than 5% in the previous month

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2015-07; Primary Completion 2017-03 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | Two weeks
  Insulin sensitivity and pancreatic response estimated with the minimal model using a frequently sampled IV glucose tolerance test

SECONDARY OUTCOMES:
Glucagon like peptide (GLP-1) change | Two weeks
  Change in fasting GLP-1 after sucralose ingestion
Ghrelin change | Two weeks
  Change in fasting ghrelin after sucralose ingestion
Tyrosine-tyrosine peptide (PYY) change | Two weeks
  Change in fasting PYY after sucralose ingestion
Leptin change | Two weeks
  Change in fasting leptin after sucralose ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Paloma Almeda-Valdes, MD, PhD, Principal Investigator — Attending Physician
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Suez J, Korem T, Zeevi D, Zilberman-Schapira G, Thaiss CA, Maza O, Israeli D, Zmora N, Gilad S, Weinberger A, Kuperman Y, Harmelin A, Kolodkin-Gal I, Shapiro H, Halpern Z, Segal E, Elinav E. Artificial sweeteners induce glucose intolerance by altering the gut microbiota. Nature. 2014 Oct 9;514(7521):181-6. doi: 10.1038/nature13793. Epub 2014 Sep 17. PMID 25231862
- [Background] Brown RJ, Walter M, Rother KI. Effects of diet soda on gut hormones in youths with diabetes. Diabetes Care. 2012 May;35(5):959-64. doi: 10.2337/dc11-2424. Epub 2012 Mar 12. PMID 22410815
- [Result] Pepino MY, Tiemann CD, Patterson BW, Wice BM, Klein S. Sucralose affects glycemic and hormonal responses to an oral glucose load. Diabetes Care. 2013 Sep;36(9):2530-5. doi: 10.2337/dc12-2221. Epub 2013 Apr 30. PMID 23633524
- [Derived] Romo-Romo A, Aguilar-Salinas CA, Brito-Cordova GX, Gomez-Diaz RA, Almeda-Valdes P. Sucralose decreases insulin sensitivity in healthy subjects: a randomized controlled trial. Am J Clin Nutr. 2018 Sep 1;108(3):485-491. doi: 10.1093/ajcn/nqy152. PMID 30535090